CLINICAL TRIAL: NCT05367505
Title: Prospective Pilot Study With a Titanium Fusion Implant in Combination With Trans-iliac Screws for Insufficiency Fractures of the Pelvis
Brief Title: Titanium Fusion Implant in Combination With Trans-iliac Screws for Insufficiency Fractures of the Pelvis
Acronym: TIKTIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: SI-BONE, Inc. (Industry); Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIKTIS
Record Dates: First submitted 2022-05-04; First posted 2022-05-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Fracture; Insufficiency Fractures; Mobility Limitation
Keywords: Fracture Fixation; Fragility Fractures; Pelvis; Surgical Procedures; Minimal Invasive
MeSH Terms: conditions — Hip Fractures; Fractures, Stress; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iFuse-3D (Experimental): Titanium fusion implant in combination with trans-iliac screws
  Interventions: Device: iFuse-3D implant

INTERVENTIONS:
Device: iFuse-3D implant — The iFuse Implant System consists of cannulated triangular titanium implants (Ti 6AI4V ELI, ASTM F136) with a porous coating of commercially pure titanium plasma spray (C.P. Ti, ASTM F1580) and a setting instrument. The coating and special shape of the implants prevent rotation or displacement of the sacroiliac (SI) joint. The placement instrument uses guide pins to achieve precise placement.

SUMMARY:
Many approaches to the surgical treatment of OF-P have been tried, but no one method has stood out as particularly successful. The placement of three implants, including implants that could minimise motion in the sacroiliac joint through early fixation and long-term fusion of the sacroiliac joint, can prevent micromotion in the fracture and thereby improve the clinical outcome of OF-Ps.

The iFuse-3D implant was shown to be safe and effective for chronic sacroiliac pain in non-osteoporotic patients.

The primary aim is to assess the proportion of patients operated on using iFuse-3D in conjunction with transiliac-transsacral screws who regain pre-fracture mobility by the time of hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Legal capacity, capacity to inform
* Presence of a written declaration of consent by the patient
* Age: ≥ 60 years
* Acute or subacute (less than 2 months) posterior pelvic girdle pain associated with low energy trauma or occurring spontaneously
* Diagnosis confirmed by CT and/or MRI
* The fracture corresponds to types OF3 and OF4 of the OF Pelvis classification.
* Prior to the fracture, there was free, non-wheelchair mobility (Functional Mobility Score of 2 or higher)

Exclusion Criteria:

* Diagnosed uncontrolled psychiatric illness (e.g. dementia, schizophrenia, major depression, personality disorder) that could affect study participation or reporting of findings
* History of pelvic fracture within one year with evidence of failure of fracture to heal or internal fixation of the pelvic ring of any type
* Patients unable to ambulate before the fracture
* Patient has had lumbar instrumentation of more than two vertebrae and/or instrumentation of S1 in the past
* Additional fractures that limit mobility
* OF-P associated with benign or malignant tumours of the pelvis
* Abnormal neurological condition that could affect study participation
* An unusual clinical condition associated with a high risk of not being able to follow up (e.g. COPD, severe heart failure, Parkinson's disease, autoimmune diseases)
* Any pelvic condition or anatomical feature that makes surgery impracticable
* Known allergy to titanium or titanium alloys
* Known opioid abuse for chronic pain syndromes
* Participation in other interventional trials
* Lack of surgical capability
* Persons in a dependent/employee relationship with the sponsor or investigator
* Placement in an institution due to court or administrative order.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who regain their pre-fracture mobility as measured by the FMS by the time of hospital discharge | Time 8 days (discharge) after surgery
  The proportion is shown with frequencies and corresponding percentages.

SECONDARY OUTCOMES:
Proportion of patients who achieve pre-fracture mobility within six weeks. | Time six weeks after surgery
  The proportion is shown with frequencies and corresponding percentages.
Proportion of patients who achieve pre-fracture mobility at three months. | Time three months after surgery
  The proportion is shown with frequencies and corresponding percentages.
Proportion of patients who achieve pre-fracture mobility at six months. | Time six months after surgery
  The proportion is shown with frequencies and corresponding percentages.
Proportion of patients who achieve pre-fracture mobility at 12 months. | Time 12 months after surgery
  The proportion is shown with frequencies and corresponding percentages.
Proportion of patients who achieved an FMS ≥ 2 (= walking with assistive devices) at discharge. | Time 8 days (discharge) after surgery
  The proportion is shown with frequencies and corresponding percentages.
Proportion of patients who achieved an FMS ≥ 2 within six weeks. | Time six weeks after surgery
  The proportion is shown with frequencies and corresponding percentages.
Proportion of patients who achieved an FMS ≥ 2 at three months. | Time three months after surgery
  The proportion is shown with frequencies and corresponding percentages.
Proportion of patients who achieved an FMS ≥ 2 at six months. | Time six months after surgery
  The proportion is shown with frequencies and corresponding percentages.
Proportion of patients who achieved an FMS ≥ 2 at 12 months. | Time 12 months after surgery
  The proportion is shown with frequencies and corresponding percentages.
Change in posterior pelvic girdle pain at rest and when attempting to walk measured by a NRS (0-10) within six weeks. | Time six weeks after surgery
  Appropriate measures of location such as medians/quartiles are calculated. Appropriate significance tests will be applied.
Change in posterior pelvic girdle pain at rest and when attempting to walk measured by a NRS (0-10) at three months. | Time three months after surgery
  Appropriate measures of location such as medians/quartiles are calculated. Appropriate significance tests will be applied.
Change in posterior pelvic girdle pain at rest and when attempting to walk measured by a NRS (0-10) at six months. | Time six months after surgery
  Appropriate measures of location such as medians/quartiles are calculated. Appropriate significance tests will be applied.
Change in posterior pelvic girdle pain at rest and when attempting to walk measured by a NRS (0-10) at 12 months. | Time 12 months after surgery
  Appropriate measures of location such as medians/quartiles are calculated. Appropriate significance tests will be applied.
Timed up and go test after six weeks. | Time six weeks after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Timed up and go test after three months. | Time three months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Timed up and go test after six months. | Time six months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Timed up and go test after 12 months. | Time 12 months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Opioid consumption and osteoporosis medication in the last six weeks. | Time six weeks after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Opioid consumption and osteoporosis medication in the last three months. | Time three months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Opioid consumption and osteoporosis medication in the last six months. | Time six months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Opioid consumption and osteoporosis medication in the last 12 months. | Time 12 months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Change in quality of life measured by the EuroQol-5D-3L after six weeks. | Time six weeks after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Change in quality of life measured by the EuroQol-5D-3L after three months. | Time three months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Change in quality of life measured by the EuroQol-5D-3L after six months. | Time six months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Change in quality of life measured by the EuroQol-5D-3L after 12 months. | Time 12 months after surgery
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. Appropriate significance tests will be applied.
Proportion of screws or iFuse fractures. | Time within 12 months
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. If necessary, appropriate significance tests are applied.
Proportion of screw sintering. | Time within 12 months
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. If necessary, appropriate significance tests are applied.
Proportion of sintering/migration of the iFuse implant. | Time within 12 months
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. If necessary, appropriate significance tests are applied.
Proportion of radiological signs of loosening. | Time within 12 months
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. If necessary, appropriate significance tests are applied.
Proportion of infections. | Time within 12 months
  Appropriate measures of location such as frequencies/percentages or medians/quartiles are calculated. If necessary, appropriate significance tests are applied.

CONTACTS AND LOCATIONS:
Overall Officials: Erol Gercek, Prof., Principal Investigator — University Medical Center of the Johannes Gutenberg University Mainz
Locations (3):
- Germany (3):
  - Diakonie Krankenhaus, Bad Kreuznach
  - University Medical Center of the Johannes Gutenberg University Mainz, Mainz
  - Helios Universitätsklinikum Wuppertal, Wuppertal

REFERENCES:
- [Background] Sullivan MP, Baldwin KD, Donegan DJ, Mehta S, Ahn J. Geriatric fractures about the hip: divergent patterns in the proximal femur, acetabulum, and pelvis. Orthopedics. 2014 Mar;37(3):151-7. doi: 10.3928/01477447-20140225-50. PMID 24762143
- [Background] Kannus P, Niemi S, Parkkari J, Sievanen H. Continuously declining incidence of hip fracture in Finland: Analysis of nationwide database in 1970-2016. Arch Gerontol Geriatr. 2018 Jul-Aug;77:64-67. doi: 10.1016/j.archger.2018.04.008. Epub 2018 Apr 17. PMID 29684740
- [Background] Kannus P, Parkkari J, Niemi S, Sievanen H. Low-Trauma Pelvic Fractures in Elderly Finns in 1970-2013. Calcif Tissue Int. 2015 Dec;97(6):577-80. doi: 10.1007/s00223-015-0056-8. Epub 2015 Aug 29. PMID 26319676
- [Background] Nanninga GL, de Leur K, Panneman MJ, van der Elst M, Hartholt KA. Increasing rates of pelvic fractures among older adults: The Netherlands, 1986-2011. Age Ageing. 2014 Sep;43(5):648-53. doi: 10.1093/ageing/aft212. Epub 2014 Jan 12. PMID 24419459
- [Background] Andrich S, Haastert B, Neuhaus E, Neidert K, Arend W, Ohmann C, Grebe J, Vogt A, Jungbluth P, Rosler G, Windolf J, Icks A. Epidemiology of Pelvic Fractures in Germany: Considerably High Incidence Rates among Older People. PLoS One. 2015 Sep 29;10(9):e0139078. doi: 10.1371/journal.pone.0139078. eCollection 2015. PMID 26418971
- [Background] Maier GS, Kolbow K, Lazovic D, Horas K, Roth KE, Seeger JB, Maus U. Risk factors for pelvic insufficiency fractures and outcome after conservative therapy. Arch Gerontol Geriatr. 2016 Nov-Dec;67:80-5. doi: 10.1016/j.archger.2016.06.020. Epub 2016 Jul 15. PMID 27448040
- [Background] Rommens PM, Wagner D, Hofmann A. Fragility Fractures of the Pelvis. JBJS Rev. 2017 Mar 21;5(3):e3. doi: 10.2106/JBJS.RVW.16.00057. No abstract available. PMID 28359073
- [Background] Breuil V, Roux CH, Carle GF. Pelvic fractures: epidemiology, consequences, and medical management. Curr Opin Rheumatol. 2016 Jul;28(4):442-7. doi: 10.1097/BOR.0000000000000293. PMID 27077891
- [Background] Pohlemann T, Stengel D, Tosounidis G, Reilmann H, Stuby F, Stockle U, Seekamp A, Schmal H, Thannheimer A, Holmenschlager F, Gansslen A, Rommens PM, Fuchs T, Baumgartel F, Marintschev I, Krischak G, Wunder S, Tscherne H, Culemann U. Survival trends and predictors of mortality in severe pelvic trauma: estimates from the German Pelvic Trauma Registry Initiative. Injury. 2011 Oct;42(10):997-1002. doi: 10.1016/j.injury.2011.03.053. Epub 2011 Apr 22. PMID 21513936
- [Background] Andrich S, Haastert B, Neuhaus E, Neidert K, Arend W, Ohmann C, Grebe J, Vogt A, Jungbluth P, Thelen S, Windolf J, Icks A. Excess Mortality After Pelvic Fractures Among Older People. J Bone Miner Res. 2017 Sep;32(9):1789-1801. doi: 10.1002/jbmr.3116. Epub 2017 May 8. PMID 28272751
- [Background] Ullrich BW, Schnake KJ, Spiegl UJA, Schenk P, Mendel T, Behr L, Bula P, Flucht LB, Franck A, Gercek E, Gruninger S, Hartung P, Jacobs C, Katscher S, Klauke F, Liepold K, Muller CW, Muller M, Osterhoff G, Partenheimer A, Piltz S, Riehle M, Sauer D, Scheyerer MJ, Schleicher P, Schmeiser G, Schmidt R, Scholz M, Siekmann H, Sprengel K, Stoevesandt D, Verheyden A, Zimmermann V; Spine Section of the German Society for Orthopaedics and Trauma. OF-Pelvis classification of osteoporotic sacral and pelvic ring fractures. BMC Musculoskelet Disord. 2021 Nov 29;22(1):992. doi: 10.1186/s12891-021-04882-6. PMID 34844577
- [Background] Hammer N, Lingslebe U, Aust G, Milani TL, Hadrich C, Steinke H. Ultimate stress and age-dependent deformation characteristics of the iliotibial tract. J Mech Behav Biomed Mater. 2012 Dec;16:81-6. doi: 10.1016/j.jmbbm.2012.04.025. Epub 2012 Oct 30. PMID 23178479